CLINICAL TRIAL: NCT00901589
Title: The Incorporation of Marine n-3 Polyunsaturated Fatty Acids in Pre- and Postmenopausal Women: a Randomized Double-Blinded Placebo-Controlled Clinical Trial
Brief Title: Marine n-3 Polyunsaturated Fatty Acids in Pre- and Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Dr., ph.d.stud. Petra Witt
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Petra Witt
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2009-05-14 (Estimated); Status verified 2009-05

CONDITIONS: Postmenopause; Premenopause
Keywords: n-3 PUFAs; menopause; adipose tissue; estrogens; Incorporation of fishoil in pre- and postmenopausal women; Marine n-3 PUFAs influence on female hormones in blood
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Premenopausal women-fishoil (Active Comparator)
  Interventions: Dietary Supplement: marine n-3 polyunsaturated fatty acids
- Premenopausal-placebo (Placebo Comparator)
  Interventions: Dietary Supplement: thistle oil
- Postmenopausal women-fishoil (Active Comparator)
  Interventions: Dietary Supplement: marine n-3 polyunsaturated fatty acids
- Postmenopausal-placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Thistle oil

INTERVENTIONS:
Dietary Supplement: marine n-3 polyunsaturated fatty acids — Four capsules daily containing 2.2 g marine n-3 polyunsaturated fatty acids in total
  Other Names: Fish oil
  Arms: Premenopausal women-fishoil
Dietary Supplement: thistle oil — four capsules a day
  Arms: Premenopausal-placebo
Dietary Supplement: marine n-3 polyunsaturated fatty acids — Four capsules daily, 2.2 g marine n-3 PUFAs in total
  Other Names: Fish oil
  Arms: Postmenopausal women-fishoil
Dietary Supplement: Thistle oil — Four capsules daily
  Arms: Postmenopausal-placebo

SUMMARY:
The study is a randomised placebo controlled double-blinded clinical trial where a group of healthy pre- and postmenopausal women is randomised to the intake of fish oil capsules or placebo oil capsules for 12 weeks. Anthropometric measurements(weight, height,blood pressure) blood samples and adipose tissue biopsies will be taken in order to illustrate the effect of marine n-3 PUFAs (fish oil) on the concentration of circulating female hormones and to investigate what impact menopause might have on the ability to incorporate marine n-3 PUFAs into tissues.

ELIGIBILITY:
Inclusion Criteria:

* age 18-70 years old
* healthy or well-treated chronic disease

Exclusion Criteria:

* hormone treatment
* foreseen compliance problem
* fish oil consumers

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Content of marine n-PUFAs as percent of total content of fatty acids in adipose tissue and in platelets before and after intervention

SECONDARY OUTCOMES:
Measurement of oestrogen concentrations in blood before and after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Center for cardiovascular research, Aalborg Hospital, Aalborg, Denmark